CLINICAL TRIAL: NCT02511639
Title: MAINtenance Afinitor: A Randomized Trial Comparing Maintenance Aromatase Inhibitors (AIs) + Everolimus (Afinitor) vs AIs in Hormone Receptor Positive (HR+) Metastatic Breast Cancer Patients With Disease Control After First Line Chemotherapy
Brief Title: Maintenance Aromatase Inhibitors (AIs)+ Everolimus vs AIs in Hormone Receptor Positive Metastatic Breast Cancer Patients
Acronym: MAIN-A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: University of Padova (Other)
Responsible Party: Principal Investigator, Pierfranco Conte, MD, PhD, Istituto Oncologico Veneto IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001JIT36T; 2013-004153-24 (EudraCT Number)
Record Dates: First submitted 2015-07-16; First posted 2015-07-30 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer Metastatic
Keywords: Hormone receptor positive; HER2 negative
MeSH Terms: interventions — Everolimus; Aromatase Inhibitors; exemestane; Letrozole; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Everolimus & Aromatase inhibitors (Experimental): Everolimus 10 mg po daily + Aromatase inhibitors (Exemestane 25 mg po daily or Letrozole 2.5 mg po daily or Anastrozole 1 mg po daily)
  Interventions: Drug: Everolimus; Drug: Aromatase Inhibitors
- Arm B: Aromatase inhibitors (Active Comparator): Aromatase inhibitors (Exemestane 25 mg po daily or Letrozole 2.5 mg po daily or Anastrozole 1 mg po daily)
  Interventions: Drug: Aromatase Inhibitors

INTERVENTIONS:
Drug: Everolimus — Everolimus is formulated as tablets of 10 mg strength for oral administration.
  Arms: Arm A: Everolimus & Aromatase inhibitors
Drug: Aromatase Inhibitors — Anastrozole is formulated as tablets of 1 mg strength for oral administration. Letrozole is formulated as tablets of 2.5 mg strength for oral administration. Exemestane is formulated as tablets of 25 mg strength for oral administration.
  Other Names: Exemestane; Letrozole; Anastrozole

SUMMARY:
The purpose of this study is to compare maintenance Aromatase Inhibitors (AIs) + everolimus with Aromatase Inhibitors alone after 1st line chemotherapy in patients with HR+ metastatic breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is:

* to compare the progression free survival (PFS) of AIs/everolimus to AIs administered as maintenance therapy in HR+ advanced breast cancer patients with disease control (Complete Response (CR), Partial Response (PR) or Stable Disease (SD))after 1st line chemotherapy.
* To evaluate the overall survival
* To assess the safety profile
* To evaluate the response rate

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old women with metastatic breast cancer
2. Histological confirmation of hormone-receptor positive (defined as at least 10% of estrogen receptor (ER) and/or progesterone receptor (PgR) positivity) and human epidermal growth factor receptor 2 (HER2) negative (score 0-1+ in immunohistochemistry or FISH negativity) breast cancer
3. Postmenopausal status
4. One line of chemotherapy for metastatic disease; patients must have received a minimum of 6 cycles of chemotherapy in order to be eligible, and must have obtained disease control (CR or PR od SD)
5. Eastern Cooperative Oncology Group (ECOG) Performance status < 2
6. Adequate bone marrow and coagulation function
7. Adequate liver function
8. Adequate renal function
9. Fasting serum cholesterol ≤ 300 mg/dl or 7.75 mmol/L and fasting triglycerides ≤ 2.5 × upper limit of normal (ULN). In case one or both of these thresholds are exceeded, the patient can only be included after initiation of statin therapy or other lipid lowering drugs (eg fibrates), and when the above mentioned values have been achieved
10. Fasting glucose < 1.5 × ULN
11. Written informed consent obtained before any screening procedure and according to local guidelines.

Exclusion Criteria:

1. HER2-overexpressing patients by local laboratory testing (immunohistochemistry 3+ staining or in situ hybridization positive)
2. Previous treatment with mammalian target of rapamycin (mTOR) inhibitors
3. Known hypersensitivity to mTOR inhibitors, e.g. sirolimus (rapamycin)
4. More than one chemotherapy line for metastatic disease
5. Treatment with angiogenetic compounds as maintenance therapy (eg. bevacizumab)
6. Radiotherapy within four weeks prior to enrollment except in case of localized radiotherapy for analgesic purpose or for lytic lesions at risk of fracture which can then be completed within two weeks prior to enrollment. Patients must have recovered from radiotherapy toxicities prior to enrollment
7. Symptomatic central nervous system metastases
8. Patients with a known history of HIV positivity
9. Active, bleeding diathesis, or on oral anti-vitamin K medication (except low dose warfarin and acetylsalicylic acid or equivalent, as long as the international normalized ratio (INR) is ≤ 2.0)
10. Any severe and / or uncontrolled medical conditions such as:

    * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to enrollment, serious uncontrolled cardiac arrhythmia
    * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 × ULN
    * Acute and chronic, active infectious disorders and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy
    * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
    * Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, diffusion capacity of lung for carbon monoxide (DLco) and O2 saturation at rest on room air should be considered to exclude restrictive pulmonary disease, pneumonitis or pulmonary infiltrates.
11. Patients who test positive for hepatitis B or C (patients who test negative for hepatitis B virus (HBV)-DNA, HBsAg, and HBcAb but positive for HBsAb with prior history of vaccination against Hepatitis B will be eligible)
12. Patients being treated with drugs recognized as being strong inhibitors or inducers of the isoenzyme Cytochrome P3A (Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itraconazole, Voriconazole, Ritonavir, Telithromycin) within the last 5 days prior to enrollment
13. History of non-compliance to medical regimens
14. Patients unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-07-30 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Up to 2 years after randomisation
  PFS is defined as the time from randomization to the first documentation of objective disease progression or death from any cause

SECONDARY OUTCOMES:
Overall survival | Up to 2 years after randomisation
  Overall survival is defined as the interval between the date of randomization and the date of patient death due to any cause, or the last date the patient was known to be alive
Response rate | Every 12 weeks during treatment, up to 2 years after randomisation
  Responses will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria only for patients with measurable disease at the time of study entry.
Safety profile | Baseline and every 4 weeks during treatment, up to 2 years after randomisation
  Toxicity will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI -CTCAE), version 4.

CONTACTS AND LOCATIONS:
Overall Officials: Pierfranco Conte, MD, PhD, Principal Investigator — Medical Oncology 2, Istituto Oncologico Veneto
Locations (16):
- Italy (16):
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti di Ancona, Ancona, AN
  - Ospedale Papa Giovanni XXIII, Bergamo, Bg
  - Policlinico Sant'Orsola Malpighi, Bologna, BO
  - ASL Brindisi "Antonio Perrini", Brindisi, BR
  - Azienda Spedali Civili di Brescia, Brescia, BS
  - A.S.O. S.Croce e Carle di Cuneo, Cuneo, CN
  - Azienda Ospedaliero - Universitaria "Policlinico - Vittorio Emanuele", Catania, CT
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna, Cona, FE
  - Ospedale Misericordia di Grosseto, Grosseto, GR
  - Istituto Nazionale dei Tumori IRCCS, Milan, MI
  - Azienda Ospedaliera Universitaria di Parma, Parma, PR
  - IRCCS - Azienda Ospedaliera S.M. Nuova, Reggio Emilia, RE
  - Ospedale Civile Santa Chiara, Trento, TN
  - Azienda Ospedaliero-Universitaria "Santa Maria della Misericordia", Udine, UD
  - Ospedale Sacro Cuore - Don Calabria, Negrar, VR
  - Ospedale dell'Angelo, Mestre

IPD SHARING:
Plan to Share IPD: No